CLINICAL TRIAL: NCT03376763
Title: MAintain the Efficacy and Safety in Treatment of Schizophrenia After Switching to Long-acTing Injectable aRipiprazole From Oral Atypical Antipsychotics
Acronym: MAESTRO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 031-402-00129
Record Dates: First submitted 2017-12-13; First posted 2017-12-18 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Schizophrenia; Antipsychotics; Long-Acting Injection; LAI; Aripiprazole
Keywords: aripiprazole; Long-Acting Injection
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Schizophrenia patients who are taking oral aripiprazole will be switched to Abilify maintena
  Interventions: Drug: Abilify maintena
- Group 2 (Experimental): Schizophrenia patients who are taking other oral atypical antipsychotics will be switched to Abilify maintena
  Interventions: Drug: Abilify maintena

INTERVENTIONS:
Drug: Abilify maintena — Switching from oral atypical antipsychotics to long-acting injectable aripiprazole (Abilify maintena)
  Other Names: long-acting injectable aripiprazole

SUMMARY:
Interventional, multicenter, open-label, 20 weeks study

* To identify efficacy and safety in switching from oral aripiprazole to Abilify Maintena.
* To identify efficacy and safety in switching from oral atypical antipsychotics other than aripiprazole to Abilify Maintena

DETAILED DESCRIPTION:
We would like to evaluate the efficacy and safety when switching to Abilify Maintena according to the approved indication of Abilify Maintena, for subjects who are taking oral antipsychotic drugs. It is expected that this will serve as a basis for suggesting a successful switching guideline from oral antipsychotics to Abilify Maintena, which can be applicable in clinical practice.

ELIGIBILITY:
Inclusion criteria

1. Subjects who voluntarily consented to participating in the clinical trial.
2. Male and female legally aged ≥19 and < 65 years.
3. Subjects who were diagnosed of schizophrenia as defined by DSM diagnostic criteria, and were diagnosed of schizophrenia for at least for 2 years prior to screening.
4. Subjects with all of the following schizophrenia clinical features:

   A. Outpatient subjects, with no hospitalization for worsening of schizophrenia within 3 months prior to screening.

   B. Subjects who have no more than a moderate rating on the PANSS total score≤80 C. 4 individual PANSS items, which are concerning to psychotic symptom (P2. conceptual disorganization, P3. hallucinatory behavior, P6. suspiciousness/persecution, G9. unusual thought content), score≤4.

   D. CGI-S score ≤4 (moderately ill).
5. Subjects who take atypical antipsychotic drugs with the therapeutic effective dose (as specified in each label) for schizophrenia treatment, and should be maintained on the type and dose of the current antipsychotic drugs (including both typical and atypical antipsychotic drugs) for at least 4 weeks prior to the screening.
6. Subjects who need antipsychotic treatment (other than clozapine), and would be stable when switching to Abilify Maintena on the investigator's judgement.
7. Subjects must exhibit willingness, physiologic capability, and an educational level sufficient to comply with all protocol procedures as per the investigator's judgment.

Exclusion criteria

1. Subject who showed medically significant adverse events or intolerance with aripiprazole during screening period or as prior experiences.
2. Subjects with a current DSM diagnostic criteria-based diagnosis other than schizophrenia, including Schizoaffective disorder, major depressive disorder, bipolar disorder, delirium, neurocognitive disorder due to Alzheimer's or similar diseases, amnesia, borderline, paranoid, histrionic, schizotypal, schizoid, antisocial or other cognitive or personality disorders.
3. Subjects with diseases of the central nervous system that may impact the assessment of the psychotic symptoms as per investigator's opinion.
4. Subjects who have been treated with clozapine, electroconvulsive therapy (ECT) or other long-acting injectable antipsychotic drugs within 3 months prior to the screening.
5. Subjects who have been treated more than 2 oral antipsychotic drugs (including both typical and atypical antipsychotic drugs) with the minimum therapeutic effective dose (as specified in each label) for schizophrenia treatment at screening.

   (e.g. Aripiprazole≥10 mg/day, Olanzapine≥10 mg/day, Risperidone≥2 mg/day, Quetiapine ≥150 mg/day)
6. Subjects who have been treated with oral antipsychotic drugs (including both typical and atypical antipsychotic drugs) exceeding maximum maintenance dose (as specified in each label) at screening.

   (e.g. Aripiprazole>30 mg/day, Olanzapine>20 mg/day, Risperidone > 6 mg/day, Quetiapine > 750 mg/day)
7. Subjects with a significant risk of violent behavior or a significant risk of committing suicide based on history or investigator's judgment.
8. Subjects had a history of seizures, neuroleptic malignant syndrome, clinically significant tardive dyskinesia, or other medical condition that would expose them to undue risk or interfere with study assessments.
9. Significant history of drug abuse disorder (excluding caffeine and nicotine, including alcohol, as defined in DSM-5 substance use disorder or in the opinion of the investigator) within the last 6 months prior to screening.
10. Subjects who participated in another interventional clinical trial within 30 days prior to screening.
11. Pregnant or lactating women, or women of childbearing potential who are not willing to or not able to use contraceptive methods (sexual abstinence; oral, implanted or injection hormone contraceptive methods; intrauterine device or condom; barrier contraceptive methods such as diaphragm and spermicide), accepted to avoid pregnancy until the end of the clinical trial.
12. Subjects having any other clinically significant finding of the physical examination or laboratory value that make investigator consider that it would be inappropriate to participate in this study.

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 201 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-19 (Actual)

PRIMARY OUTCOMES:
PANSS total score | 16 weeks
  Change in PANSS total score from baseline to Week 16

SECONDARY OUTCOMES:
CGI-S | 16 weeks
  Change in CGI-S (severity) from baseline to Week 16
CGI-I | 16 weeks
  Mean CGI-I (improvement) score at Week 16
PANSS positive and negative subscale score | 16 weeks
  Change in PANSS positive and negative subscale score from baseline to Week 16
IAQ score | 16 weeks
  Mean IAQ score at Week 16

OTHER OUTCOMES:
study discontinuation rates | 16 weeks
  Comparison the study discontinuation rates between Group 1 and Group 2
study discontinuation rates | 16 weeks
  Comparison the study discontinuation rates in Group 2 depending on the other oral atypical antipsychotics
proportion of subjects who have more than 20% increased rating on the PANSS total score | 16 weeks
  Comparison the proportion of subjects who have more than 20% increased rating on the PANSS total score from baseline to Week 16 between Group 1and Group 2
proportion of subjects who have more than 20% increased rating on the PANSS total score | 16 weeks
  Comparison the proportion of subjects who have more than 20% increased rating on the PANSS total score from baseline to Week 16 in Group 2 depending on the other oral atypical antipsychotics

CONTACTS AND LOCATIONS:
Overall Officials: Jun Soo Kwon, Dr., Principal Investigator — Seoul National University Hospital
Locations (27):
- South Korea (27):
  - Gongju National Hospital, Gongju, Chungcheongnam-do
  - Hanyang University Guri Hospital, Guri-si, Gyeonggi-do
  - Cha Bundang Medical Center, Seongnam-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - The Catholic University of Korea Uijeongbu ST. Mary'S Hospital, Uijeongbu-si, Gyeonggi-do
  - Yong-In Mental Hospital, Yongin-si, Gyeonggi-do
  - Jeju National University Hospital, Jeju City, Jeju-do
  - Chonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Konkuk University Chungju Hospital, Chungju, North Chungcheong
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National University Hospital, Daegu
  - Yeungnam University Medical Center, Daegu
  - Eulji University Hospital, Daejeon
  - Konyang University Hospital, Daejeon
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Inha University Hospital, Incheon
  - International St. Mary's Hospital, Incheon
  - Inje University Haeundae Paik Hospital, Pusan
  - Pusan National University Yangsan Hospital, Pusan
  - Kangbuk Samsung Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Eulji General Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Kyung Hee University Hospital, Seoul
  - Seoul National University Hosipital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aripiprazole Investigator Brochure, Version No. 20, 16 Aug 2016
- [Result] Regier DA, Narrow WE, Rae DS, Manderscheid RW, Locke BZ, Goodwin FK. The de facto US mental and addictive disorders service system. Epidemiologic catchment area prospective 1-year prevalence rates of disorders and services. Arch Gen Psychiatry. 1993 Feb;50(2):85-94. doi: 10.1001/archpsyc.1993.01820140007001. PMID 8427558
- [Result] Hong Kyu Ihm et al. Factors Related to Medication Adherence in Outpatients with Schizophrenia under More Than 5 Years of Treatment. J Korean Neuropsychiatr Assoc 2016; 55(4):397-406
- [Result] Hyun-Ku Kang, et al. Safety and Effectiveness of Long Acting Injectable Antipsychotic Paliperidone Palmitate Treatment in Schizophrenics: A 24-Week Open-Label Study. Korean J Biol Psychiatry 2013;20:111-117
- [Result] Gilbert PL, Harris MJ, McAdams LA, Jeste DV. Neuroleptic withdrawal in schizophrenic patients. A review of the literature. Arch Gen Psychiatry. 1995 Mar;52(3):173-88. doi: 10.1001/archpsyc.1995.03950150005001. No abstract available. PMID 7872841
- [Result] Gitlin M, Nuechterlein K, Subotnik KL, Ventura J, Mintz J, Fogelson DL, Bartzokis G, Aravagiri M. Clinical outcome following neuroleptic discontinuation in patients with remitted recent-onset schizophrenia. Am J Psychiatry. 2001 Nov;158(11):1835-42. doi: 10.1176/appi.ajp.158.11.1835. PMID 11691689
- [Result] Kane JM, Sanchez R, Perry PP, Jin N, Johnson BR, Forbes RA, McQuade RD, Carson WH, Fleischhacker WW. Aripiprazole intramuscular depot as maintenance treatment in patients with schizophrenia: a 52-week, multicenter, randomized, double-blind, placebo-controlled study. J Clin Psychiatry. 2012 May;73(5):617-24. doi: 10.4088/JCP.11m07530. PMID 22697189
- [Result] Naber D, Hansen K, Forray C, Baker RA, Sapin C, Beillat M, Peters-Strickland T, Nylander AG, Hertel P, Andersen HS, Eramo A, Loze JY, Potkin SG. Qualify: a randomized head-to-head study of aripiprazole once-monthly and paliperidone palmitate in the treatment of schizophrenia. Schizophr Res. 2015 Oct;168(1-2):498-504. doi: 10.1016/j.schres.2015.07.007. Epub 2015 Jul 29. PMID 26232241
- [Result] Seockhoon Chung, Chang Yoon Kim. et al. Effectiveness and Tolerability of Long-Acting Risperidone：A 12 Weeks, Multi-center Switching Study from Oral Antipsychotics. Korean J Psychopharmacol 16/2:109-120, 2005
- [Result] Fleischhacker WW, Sanchez R, Perry PP, Jin N, Peters-Strickland T, Johnson BR, Baker RA, Eramo A, McQuade RD, Carson WH, Walling D, Kane JM. Aripiprazole once-monthly for treatment of schizophrenia: double-blind, randomised, non-inferiority study. Br J Psychiatry. 2014 Aug;205(2):135-44. doi: 10.1192/bjp.bp.113.134213. Epub 2014 Jun 12. PMID 24925984
- See also: Clinical trial guideline for Antipsychotics; Ministry Food And Drug, 2015.09. — http://mfds.go.kr/index.do?mid=1769&seq=12790
- See also: The survey of Mental Disorders in Korea; Ministry of Health and Welfare, 2016 — http://www.korea.kr/archive/expDocView.do?docId=37547